CLINICAL TRIAL: NCT07347964
Title: The Effect of Sleep Hygiene Education on Sleep Quality and Glycemic Control in Patients With Type 2 Diabetes
Brief Title: Sleep Hygiene Education in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Oğulcan Çöme, Doctor, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/18-18
Record Dates: First submitted 2025-12-20; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes Mellitus and the Effect of Sleep Hygiene Education on Sleep Quality and Glycemic Control
Keywords: Type 2 Diabetes Mellitus; Sleep Hygiene Education; Sleep Quality; Glycemic Control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Usual Care (No Intervention): Participants in the control arm receive usual care without any structured sleep hygiene education intervention. They continue their routine diabetes management and follow-up as provided in standard clinical practice. No additional behavioral or educational intervention related to sleep is administered during the study period.
- İntervention (Experimental): Participants in this arm receive a structured sleep hygiene education program in addition to usual diabetes care. The education includes guidance on sleep-wake routines, sleep environment optimization, caffeine and screen use reduction, and behavioral strategies to improve sleep quality. The intervention is delivered through standardized educational sessions and written materials
  Interventions: Behavioral: Sleep Hygiene Education

INTERVENTIONS:
Behavioral: Sleep Hygiene Education — Participants in this arm receive a structured sleep hygiene education program in addition to usual diabetes care. The education includes guidance on sleep-wake routines, sleep environment optimization, caffeine and screen use reduction, and behavioral strategies to improve sleep quality. The intervention is delivered through standardized educational sessions and written materials.
  Arms: İntervention

SUMMARY:
The aim of this study is to evaluate the effect of sleep hygiene education on sleep quality and glycemic control of Type 2 Diabetes patients. Patients between the ages of 18-65, who were registered to the Gaziemir 11 No. Dokuz Eylül Education Family Health Centers and applied to the polyclinic, and had Type 2 Diabetes diagnosis for at least 1 year were included in the study. In the patient group in which the study will be conducted, the patients who will be applied the Pittsburgh Sleep Quality Index (PSQI) and those with a PSQI score of more than 5 were included in the study. A sociodemographic questionnaire was applied to the participants, the last measured HbA1c values were questioned, and fingertip fasting blood sugars were measured. Sleep hygiene training was applied to the intervention group at the first admission, a sleep hygiene rules checklist was given and they were asked to keep a two-week sleep diary. After the two-week sleep diary, the participants in the intervention group were given training on these issues by determining the things that could impair the quality of their sleep through the sleep diary they kept. Sleep training and sleep hygiene rules checklist were given to the control group after three months of follow-up. At the end of the 3-month follow-up, PSQI was applied to both groups again, and the last measured HbA1c values were recorded and fingertip fasting blood glucose was measured.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus for at least 1 year
* Aged 18-65 years
* Pittsburgh Sleep Quality Index (PSQI) score > 5

Exclusion Criteria:

* Use of sedative medications
* Working night shifts
* Receiving pharmacological or non-pharmacological treatment for a diagnosed -sleep disorder
* Dementia or psychiatric disorder due to an organic or general medical condition, or history of psychotic disorder or bipolar disorder
* Pregnancy
* Change in diet or diabetes treatment regimen during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Change in Sleep Quality (Pittsburgh Sleep Quality Index, PSQI) | 3 Months
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The primary endpoint is the change in PSQI total score from baseline to post-intervention (end of follow-up), with lower scores indicating better sleep quality.

SECONDARY OUTCOMES:
Change in Glycemic Control (HbA1c) | 3 Months
  Glycemic control will be assessed using glycated hemoglobin (HbA1c, %). The secondary outcome is the change in HbA1c levels from baseline to post-intervention (end of follow-up).

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be shared publicly due to ethical concerns. Data may be made available upon reasonable request, subject to approval by the ethics committee and in accordance with data protection regulations.